CLINICAL TRIAL: NCT00997191
Title: Intravitreal Bevacizumab and Intravitreal Triamcinolone Associated to Laser Photocoagulation for Diabetic Macular Edema(IBeTA)
Brief Title: Intravitreal Bevacizumab and Triamcinolone Associated to Laser Photocoagulation for Diabetic Macular Edema(IBeTA)
Acronym: IBeTA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Rodrigo Jorge, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6826/2009
Record Dates: First submitted 2009-10-15; First posted 2009-10-19 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-02

CONDITIONS: Diabetic Macular Edema
Keywords: Bevacizumab; Diabetes; Intravitreal; Macular edema; triamcinolone; VEGF
MeSH Terms: conditions — Diabetes Mellitus; Macular Edema | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Laser Group (Active Comparator): Focal / grid Laser photocoagulation in diabetic macular edema
  Interventions: Procedure: Laser photocoagulation
- Triamcinolone group (Experimental): Intravitreal triamcinolone associated to laser photocoagulation for diabetic macular edema
  Interventions: Drug: Intravitreal triamcinolone
- Bevacizumab group (Experimental): Intravitreal Bevacizumab associated to laser photocoagulation for diabetic macular edema
  Interventions: Drug: Intravitreal bevacizumab

INTERVENTIONS:
Procedure: Laser photocoagulation — Focal / grid photocoagulation for diabetic macular edema according to ETDRS guidelines
  Arms: Laser Group
Drug: Intravitreal triamcinolone — Intravitreal preservative-free triamcinolone (4mg) associated to focal photocoagulation for diabetic macular edema on baseline; Re-treatment at weeks 20 and 40 if CMT>275um
  Other Names: Triancinolona (Ophthalmos)
  Arms: Triamcinolone group
Drug: Intravitreal bevacizumab — Intravitreal bevacizumab (1.5mg) associated to focal photocoagulation for diabetic macular edema at baseline; Re-treatment at weeks 20 and 40 if CMT>275um
  Other Names: Avastin
  Arms: Bevacizumab group

SUMMARY:
Intravitreal triamcinolone has been effective for central macular thickness reduction and concomitant visual acuity improvement in patients with diabetic macular edema (DME). VEGF is a very effective inducer of permeability, being 50.000 times more potent than histamine, and may exert its effect on retinal vascular permeability by altering tight-junctions proteins, such as occluding and VE-cadherin. Based on these principles, there is a rationale for anti-VEGF agents treatment of increased retinal capillary permeability conditions, such as diabetic macular edema. Therefore, the purpose of this study is to evaluate the effects of intravitreal bevacizumab and intravitreal triamcinolone associated to laser photocoagulation for diabetic macular edema.

DETAILED DESCRIPTION:
Macular edema is a leading cause of decreased visual acuity in patients with diabetic retinopathy1,2.

Laser photocoagulation is the standard of care treatment for diabetic macular edema, based on ETDRS and recent clinical trials findings3,4. However, because visual acuity improvement post-laser is observed infrequently, and because of the frequent recurrence or persistence of DME (refractory DME) after appropriate laser treatment, particularly in eyes presenting with angiographically diffuse macular edema5-9, there is a need for alternative treatments for the management of DME. In addition, for some patients with significant cataract, precise visualization of posterior pole structures may not be possible, so that pharmacological therapy with intravitreal agents may be preferable over laser treatment.

Recent studies have shown promising results of pharmacological therapies for Diabetic macular edema. Triamcinolone has shown similar results when compared to ranibizumab and deferred focal/grid LASER in pseudophakic eyes (DRCRnet, prompt versus deferred). Ranibizumab associated with deferred LASER or as monotherapy has also shown promising results (RISE and RIDE). However, there are several concerns regarding long-term intravitreal injections therapies that include economic feasibility for the public health system, risk of endophthalmitis and patient acceptability. For these reasons, the present study decided to check associations between LASER and drug therapy, in an attempt to improve focal/grid laser outcomes with reduced number of intravitreal injections.

ELIGIBILITY:
Inclusion Criteria:

* Clinically significant DME - by biomicroscopic evaluation with generalized breakdown of the inner blood-retina barrier with diffuse fluorescein leakage involving the foveal center and most of the macular area on fluorescein angiography
* Snellen logarithm of minimum angle of 20/40 or worse
* Central macular thickness greater than 275 µm on optical coherence tomography (OCT)

Exclusion Criteria:

* Glycosylated hemoglobin rate above 10%
* History of glaucoma or ocular hypertension
* Systemic corticoid therapy
* History of thromboembolic event (including myocardial infarction or cerebral vascular accident)
* Major surgery within the prior 6 months or planned within the next 28 days
* Uncontrolled hypertension
* Severe systemic disease
* Any condition affecting documentation or follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Best Corrected Visual acuity | One Year

SECONDARY OUTCOMES:
Macular Mapping Test | One Year
Multifocal Electroretinogram | One Year
Central Macular Thickness | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Maria L Paccola, MD, Study Chair — HC FMRP - USP; André M V Messias, PhD, Study Chair — HCFMRP - USP; Bianka Y N Y Katayama, MD, Study Director — HC FMRP - USP; Rodrigo Jorge, PhD, Principal Investigator — HC FMRP - USP; Rogério A Costa, PhD, Study Chair — HC FMRP - USP
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Background] Paccola L, Costa RA, Folgosa MS, Barbosa JC, Scott IU, Jorge R. Intravitreal triamcinolone versus bevacizumab for treatment of refractory diabetic macular oedema (IBEME study). Br J Ophthalmol. 2008 Jan;92(1):76-80. doi: 10.1136/bjo.2007.129122. Epub 2007 Oct 26. PMID 17965109
- [Background] Bonini-Filho MA, Jorge R, Barbosa JC, Calucci D, Cardillo JA, Costa RA. Intravitreal injection versus sub-Tenon's infusion of triamcinolone acetonide for refractory diabetic macular edema: a randomized clinical trial. Invest Ophthalmol Vis Sci. 2005 Oct;46(10):3845-9. doi: 10.1167/iovs.05-0297. PMID 16186372
- [Background] Photocoagulation for diabetic macular edema. Early Treatment Diabetic Retinopathy Study report number 1. Early Treatment Diabetic Retinopathy Study research group. Arch Ophthalmol. 1985 Dec;103(12):1796-806. PMID 2866759
- [Background] Garner A. Pathology of diabetic retinopathy. Br Med Bull. 1970 May;26(2):137-42. doi: 10.1093/oxfordjournals.bmb.a070765. No abstract available. PMID 4192644
- [Background] Early photocoagulation for diabetic retinopathy. ETDRS report number 9. Early Treatment Diabetic Retinopathy Study Research Group. Ophthalmology. 1991 May;98(5 Suppl):766-85. PMID 2062512
- [Background] Jorge R, Costa RA, Calucci D, Cintra LP, Scott IU. Intravitreal bevacizumab (Avastin) for persistent new vessels in diabetic retinopathy (IBEPE study). Retina. 2006 Nov-Dec;26(9):1006-13. doi: 10.1097/01.iae.0000246884.76018.63. PMID 17151487
- [Background] Jonas JB, Kreissig I, Sofker A, Degenring RF. Intravitreal injection of triamcinolone for diffuse diabetic macular edema. Arch Ophthalmol. 2003 Jan;121(1):57-61. PMID 12523885
- [Background] Lee CM, Olk RJ. Modified grid laser photocoagulation for diffuse diabetic macular edema. Long-term visual results. Ophthalmology. 1991 Oct;98(10):1594-602. doi: 10.1016/s0161-6420(91)32082-7. PMID 1961650
- [Background] Kang SW, Sa HS, Cho HY, Kim JI. Macular grid photocoagulation after intravitreal triamcinolone acetonide for diffuse diabetic macular edema. Arch Ophthalmol. 2006 May;124(5):653-8. doi: 10.1001/archopht.124.5.653. PMID 16682586
- [Background] Karacorlu M, Ozdemir H, Senturk F, Arf Karacorlu S, Uysal O. Macular function by multifocal electroretinogram in diabetic macular edema after intravitreal triamcinolone acetonide injection. Eur J Ophthalmol. 2008 Jul-Aug;18(4):601-8. doi: 10.1177/112067210801800417. PMID 18609482
- [Background] Martidis A, Duker JS, Greenberg PB, Rogers AH, Puliafito CA, Reichel E, Baumal C. Intravitreal triamcinolone for refractory diabetic macular edema. Ophthalmology. 2002 May;109(5):920-7. doi: 10.1016/s0161-6420(02)00975-2. PMID 11986098
- [Background] Kook D, Wolf A, Kreutzer T, Neubauer A, Strauss R, Ulbig M, Kampik A, Haritoglou C. Long-term effect of intravitreal bevacizumab (avastin) in patients with chronic diffuse diabetic macular edema. Retina. 2008 Oct;28(8):1053-60. doi: 10.1097/IAE.0b013e318176de48. PMID 18779710
- [Background] Larsson J, Zhu M, Sutter F, Gillies MC. Relation between reduction of foveal thickness and visual acuity in diabetic macular edema treated with intravitreal triamcinolone. Am J Ophthalmol. 2005 May;139(5):802-6. doi: 10.1016/j.ajo.2004.12.054. PMID 15860283
- [Background] Soheilian M, Ramezani A, Bijanzadeh B, Yaseri M, Ahmadieh H, Dehghan MH, Azarmina M, Moradian S, Tabatabaei H, Peyman GA. Intravitreal bevacizumab (avastin) injection alone or combined with triamcinolone versus macular photocoagulation as primary treatment of diabetic macular edema. Retina. 2007 Nov-Dec;27(9):1187-95. doi: 10.1097/IAE.0b013e31815ec261. PMID 18046223
- [Background] Vujosevic S, Pilotto E, Bottega E, Benetti E, Cavarzeran F, Midena E. Retinal fixation impairment in diabetic macular edema. Retina. 2008 Nov-Dec;28(10):1443-50. doi: 10.1097/IAE.0b013e318183571e. PMID 18997608